CLINICAL TRIAL: NCT02467283
Title: Gene Expression Profiles in Chronic Periodontitis: A Gene Network-based Microarray Analysis
Brief Title: Gene Expression Profiles in Chronic Periodontitis
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Esra Guzeldemir-Akcakanat, Associate Profesor, Kocaeli University
Other Study IDs: KOU KAEK 2013 / 15
Record Dates: First submitted 2015-06-03; First posted 2015-06-10 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Chronic Periodontitis
Keywords: chronic periodontitis; genetics; microarray analysis; gingiva; genes; inflammation
MeSH Terms: conditions — Chronic Periodontitis; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Chronic Periodontitis: All subjects were free of systemic diseases and to be included, individuals had to be older than 18 years of age.
  Chronic periodontitis was diagnosed according to American Academy of Periodontology 1999 Consensus Report.
  Interventions: Genetic: Genom-based whole-genome transcriptomic
- Control Patients: Control subjects had no radiographic evidence of bone loss or any sign of past and present periodontitis.
  All subjects were free of systemic diseases and to be included, individuals had to be older than 18 years of age.
  Interventions: Genetic: Genom-based whole-genome transcriptomic

INTERVENTIONS:
Genetic: Genom-based whole-genome transcriptomic — Gene expression profiling is a powerful means of generating comprehensive genome-level data sets.

SUMMARY:
Current concepts of the causes of periodontitis implicate a bacterial infection as the primary cause of the disease. Several bacterial species residing in a biofilm on tooth surfaces are closely associated with periodontitis. Chronic periodontitis (CP) is initiated and sustained by bacterial plaque, but host defense mechanisms play an integral role in its pathogenesis.

Gene expression profiling is a powerful means of generating comprehensive genome-level data sets on diseases such as cancer, asthma, rheumatoid disorders and periodontitis, and provides significant insight information for these diseases. Gene expression profiling may provide an evidence for involving genes in the pathogenesis of CP and generate further information other than clinical signs and symptoms of CP.

The aim of this study was to identify gene-expression patterns of patients with chronic periodontitis by whole-transcriptome gene-expression analyses.

ELIGIBILITY:
Inclusion Criteria:

1. CP patients had at least 20 teeth exhibiting >30% of measured sites with >5mm clinical attachment loss.
2. Had bleeding on probing (BOP) at >50% of the proximal sites.

Exclusion Criteria:

1. Had any known systemic diseases that can influence the periodontal status, oral diseases other than chronic periodontitis and ongoing orthodontic therapy.
2. History of hepatitis, HIV infection, or diabetes; requirement for antibiotic prophylaxis, pregnancy or lactation; and long-term use of anti-inflammatory drugs.
3. Should be free of systemic diseases
4. Individuals had to be older than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patientswere recruited from those patients seeking dental treatment in Kocaeli University, Faculty of Dentistry Periodontology Clinics.
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
mRNA quantification | 2 months

SECONDARY OUTCOMES:
Gen networking map | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Esra Guzeldemir-Akcakanat, DDS, PhD, Principal Investigator — Chair and Associate Professor of Dept. of Periodontology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armitage GC. Development of a classification system for periodontal diseases and conditions. Ann Periodontol. 1999 Dec;4(1):1-6. doi: 10.1902/annals.1999.4.1.1. PMID 10863370
- [Background] Demmer RT, Behle JH, Wolf DL, Handfield M, Kebschull M, Celenti R, Pavlidis P, Papapanou PN. Transcriptomes in healthy and diseased gingival tissues. J Periodontol. 2008 Nov;79(11):2112-24. doi: 10.1902/jop.2008.080139. PMID 18980520
- [Background] Savli H, Sunnetci D, Cine N, Gluzman DF, Zavelevich MP, Sklyarenko LM, Nadgornaya VA, Koval SV. Gene expression profiling of B-CLL in Ukrainian patients in post-Chernobyl period. Exp Oncol. 2012;34(1):57-63. PMID 22453151